CLINICAL TRIAL: NCT02820272
Title: Cold Water for Reducing Pain in Negative Pressure Wound Therapy Dressing Change
Brief Title: Water for Reducing Pain in Negative Pressure Wound Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Apichai Angspatt, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 344/55
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Treatment
Keywords: Cold water; Negative pressure wound therapy; pain
MeSH Terms: conditions — Pain | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NPWT with cold water (Experimental): Each patient will be randomized for dressing method sequence, and each of them would be treated for total of three times of NPWT dressing changes over study period. This arm was the intervention with injection of cold sterile water kept in 4°C temperature into sponge 10 minutes before dressing change.
  Interventions: Procedure: NPWT with cold water
- NPWT with normal saline room temp (Active Comparator): Each patient will be randomized for dressing method sequence, and each of them would be treated for total of three times of NPWT dressing changes over study period. This arm was the intervention with injection of room temperature sterile water kept in room temperature into sponge 10 minutes before dressing change.
  Interventions: Procedure: NPWT with normal saline room temp
- NPWT without other intervention (Placebo Comparator): Each patient will be randomized for dressing method sequence, and each of them would be treated for total of three times of NPWT dressing changes over study period. This arm was no injection of any liquids into sponge before dressing change.
  Interventions: Procedure: NPWT without other intervention

INTERVENTIONS:
Procedure: NPWT with cold water — Each of dressing change would be treated with NPWT and injection of cold sterile water kept in 4°C temperature into sponge 10 minutes before dressing change
  Arms: NPWT with cold water
Procedure: NPWT with normal saline room temp — Each of dressing change would be treated with NPWT and injection of room temperature sterile water kept in room temperature into sponge 10 minutes before dressing change
  Arms: NPWT with normal saline room temp
Procedure: NPWT without other intervention — Each of dressing change would be treated with NPWT without injection of any liquids into sponge before dressing change
  Arms: NPWT without other intervention

SUMMARY:
Negative pressure wound therapy (NPWT) is a technique using vacuum dressing to promote wound healing in complicated wound. However for many patients, the application and removal of the NPWT is source of procedural pain. Some techniques had been reported to reduce these pain such as administering topical lidocain or normal saline solution before the dressing change. The authors hypothesized that administering cold water into the NPWT sponge would decrease pain during dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* Open wounded patient who is treated by negative pressure wound therapy (NPWT) with the age between 18-70 years old.

Exclusion Criteria:

* The patient who has decrease sensation at cured wound region
* The patient who has Glasgow coma scale less than 15
* The patient who cannot provide pain scale data
* The patient who has diabetic ulcer or other chronic sores
* The patient who denies to participate in research project.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain reduction during dressing changes assessed by Visual Analogue Scale (VAS) | 3 days

REFERENCES:
- [Derived] Fernandez R, Green HL, Griffiths R, Atkinson RA, Ellwood LJ. Water for wound cleansing. Cochrane Database Syst Rev. 2022 Sep 14;9(9):CD003861. doi: 10.1002/14651858.CD003861.pub4. PMID 36103365